CLINICAL TRIAL: NCT01114243
Title: Pilot Study: Ultrasound Assessment of Steroid Joint Injections in Juvenile Idiopathic Arthritis
Brief Title: Ultrasound Assessment of Steroid Joint Injections in Juvenile Idiopathic Arthritis
Status: Withdrawn | Type: Observational
Why Stopped: The PI has left Stanford University.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SU-03112010-5202; IRB Protocol 17660
Record Dates: First submitted 2010-03-30; First posted 2010-05-03 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrasound imaging

SUMMARY:
Juvenile idiopathic arthritis (JIA) is a serious autoimmune childhood disease that encompasses several types of chronic arthritis. It is the most common rheumatic disease in children and can cause significant short-term and long-term disability, including permanent joint damage. Management of JIA is based on a combination of pharmacologic interventions, physical and occupational therapy, and psychosocial support. Intra-articular steroid (IAS) injection, or injection of steroid medication into an arthritic joint, is a routine therapeutic procedure in clinical rheumatology. Most pediatric rheumatologists currently perform injections based on knowledge of anatomy and by feeling for anatomical landmarks, but results from adult studies on ultrasound (US)-guided technique have suggested a role for using US in treating and managing JIA. The overall goal of this project is to determine the feasibility of a multicenter study comparing US-guided IAS injection with the usual technique of using external anatomic features to improve arthritis symptoms in JIA. The key issues that this pilot project will determine will be: 1) the ability to use US to successfully image and detect abnormalities in the joints in children with JIA 2) image the injected medication in the joint space or its surroundings immediately after the injection 3) determine methods to measure the clinical response to injection 4) evaluate the feasibility of using saved US scans to localize injected medication in or around the joints and to determine abnormalities concerning for arthritis. These results will be used to establish the protocols necessary to design a multicenter study to determine the effect of US-guided IAS injection in the treatment of juvenile arthritis. Studies regarding the applicability and feasibility of musculoskeletal US in an outpatient pediatric rheumatology setting are important in order to establish the utility of this new technology in guiding diagnosis and therapy in JIA. Results from this study may have a significant impact on pediatric rheumatology and the way by which pediatric rheumatologists currently assess signs of arthritis and perform routine therapeutic procedures.

DETAILED DESCRIPTION:
AIM 1: The first aim will be a two-part cross-sectional study comparing US imaging of active joints in 55 subjects with JIA to standardized clinical and functional measures, assuming that each subject will have at least 1 active joint. Subjects less than 21 years diagnosed with JIA per classification described by the International League Against Rheumatism (ILAR) with large and medium joint synovitis will be eligible.

* Phase 1. A pediatric rheumatologist will examine 25 subjects with a spectrum of arthritis severity after informed consent is obtained. Large and medium joints, such as knees, ankles, wrists, and elbows, will be assessed for active arthritis, as defined by swelling or limitation of motion with pain or warmth. Grading of clinical severity is derived from the ACR Pediatric 30 and will assess for swelling on a scale of 0-3 and limitation of motion with warmth or pain on motion on a scale of 0-3. Based on this grading, a Clinical Severity Score for inactive, mild, moderate, or severe arthritis will be obtained for each joint. Following the clinical evaluation, a pediatric rheumatologist who has received training in musculoskeletal US (PI) will image the joint. A portable US machine with a high frequency probe (6-18 MHz) and power Doppler capability will be used to image the target joints and to identify anatomical signs suggestive of arthritis. At least 2 views, coronal and transverse, of each joint will be obtained and recorded per musculoskeletal US specifications as described by the European League Against Rheumatism (EULAR). US images will be saved under a subject code on the US machine hard drive. These images will be reviewed with a consulting rheumatologist with expertise in musculoskeletal US (J. Nishio, MD). US determination of synovitis (synovial thickness with Doppler enhancement), effusion, erosions, and tenosynovitis will be based on definitions established by the Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) 7 consensus group for adults with rheumatologic disease. An US score for arthritis will then be developed based on the gold standard of clinical exam. The US score will assess for active arthritis as defined by synovitis on a scale of 0-3 and/or effusion on a scale of 0-3. In addition, other significant abnormalities in the joints will be evaluated, including absence or presence of erosions and tenosynovitis. The result of this phase of Aim 1 will be the creation of an US Severity Score for inactive, mild, moderate, or severe arthritis in a single large or medium joint that is consistent with the Clinical Severity Score.
* Phase II. The US Severity Score developed as described above will be tested for correlation with the Clinical Severity Score. An additional 30 subjects meeting inclusion criteria will be enrolled and assessed for arthritis by physical exam performed by a pediatric rheumatologist followed by an US exam performed by the PI. If the subject has more than 1 large or medium joint with arthritis, a single joint will be chosen by random selection. Based on the findings, the clinician will assign a clinical score, and the PI and the consulting rheumatologist will assign an US score based on the standardized US Severity Score obtained from Phase I. The PI and consulting rheumatologist will be masked to physical exam findings and the Clinical Severity Score. The US score will then be compared to the clinical score to assess how the US scoring relates with the standardized clinical measures.

AIM 2: The second aim will study the use of US in imaging the placement of IAS and response to this therapy in 20 subjects receiving IAS for treatment of active arthritis in large and medium joints. Patients less than 21 years old with a diagnosis of JIA per ILAR classification receiving IAS injections of the knee, wrist, elbow, or ankle as part of their standard medical care will be eligible. Non-eligible patients include subjects with a non-inflammatory diagnosis, such as mechanical joint disease, or a large joint effusion requiring additional therapeutic procedures, such as arthrocentesis. Informed consent and assent for children over 7 will be obtained. The targeted joint will be scored by a rheumatologist other than the PI using the Clinical Severity Score described above. Sedation may be provided per routine for joint injection. Routine process for joint injection will be followed. The pediatric rheumatologist performing the injection will use standard external clinical landmarks and palpation to identify the appropriate injection site. Triamcinolone hexacetonide with 1% unbuffered lidocaine will then be shaken to allow the introduction of air per GAS-graphy technique as described by Koski et al. and injected into the targeted joint. The PI, who will not perform any injections in this study, will obtain US imaging just prior and immediately following the joint injection. The rheumatologist performing the injection will be masked to US images. Each image will be obtained and recorded using EULAR specifications, saved under a subject code on the US machine hard drive, and scored by the PI and the consulting rheumatologist using the US Severity Score described above. For the second aim, I will also determine the presence or absence of steroid within the target joint capsule. The physician performing the physical exam, the subject, and the subject's guardian(s) will be masked regarding US results, including location of steroid within or around the joint space and sonographic recordings of joint pathology. Patient outcomes will be determined at 1 week, 4-6 weeks and 3-6 months by the Clinical Severity Score and by US using the US Severity Score described and developed in Aim 1. The clinician performing the physical exam and the sonographer will be masked to each other's scores.

Other variables will also be collected as part of both aims, including pain as assessed by a standardized pain scale, physician assessment of global disease activity, and functional status as determined by the childhood health assessment questionnaire (CHAQ), a validated, reliable measure of functional status in JIA. These last assessments are 3 of the 6 measures of the ACR Pediatric 30, a validated measure used in clinical trials in JIA (Giannini et al., 1997). Other patient data that will be collected include JIA subtype, duration of disease, age of onset, age at procedure, race/ethnicity, concurrent medications, and whether the procedure required the use of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:The first aim will be a two-part cross-sectional study comparing US imaging of active joints in 55 subjects with JIA to standardized clinical and functional measures, assuming that each subject will have at least 1 active joint. All subjects must meet the following criteria

* Less than 21 years old
* Have a diagnosis of JIA per ILAR classification
* Have large and/ or medium joint synovitis

The second aim will study the use of US in imaging the placement of IAS and response to this therapy in 20 subjects receiving IAS for treatment of active arthritis in large and medium joints. Subjects must meet the following criteria:

* Less than 21 years old
* Have a diagnosis of JIA per ILAR classification
* Will be receiving IAS injections of the knee, wrist, elbow, and/or ankle as part of their standard medical care Exclusion Criteria:- Subjects with a non-inflammatory diagnosis, such as mechanical joint disease
* Subjects with a large joint effusion requiring additional therapeutic procedures, such as arthrocentesis
* Subjects 21 years old or older
* Subjects without a diagnosis of JIA per ILAR classification
* Subjects without large and/or medium joint synovitis
* Subjects who do not require IAS injections of the knee, wrist, elbow, and/or ankle as part of standard medical care (for Aim 2 subjects)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will enroll any gender and/or ethnic background child or young adult meeting the inclusion/exclusion criteria as detailed above.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Steroid within the joint vs out of the joint | Within 15 minutes of joint injection
Each joint will receive a Clinical Score assessing swelling and limitation of motion with warmth or pain on motion on a scale of 0-3. Each joint will also receive an US Score which will assess effusion and/or synovitis on a scale of 0-3. | 6 months to 1 year

SECONDARY OUTCOMES:
Changes in arthritis after steroid injection as defined by changes in clinical scoring and ultrasound scoring using Clinical Severity Score and Ultrasound Severity Score as defined above. | 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Christy I. Sandborg, Principal Investigator — Stanford University; Johanna Chi Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States